CLINICAL TRIAL: NCT05500469
Title: Endothelial Cell Loss in Pseudophakic Patients Receiving a Paul Glaucoma Drainage Device With Its Tube Inserted in the Anterior Versus Posterior Chamber: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oogziekenhuis Rotterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OZR-2022-03; NL81305.078.22 (Other: CCMO); MEC-2022-0364 (Other: MEC)
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDD-tube in anterior chamber (Active Comparator): The Paul glaucoma drainage device consists of a plate and a tube. During surgery the plate is positioned underneath the conjunctiva and two extraocular muscles in the upper temporal or nasal quadrant of the eye. The tube is positioned in the anterior chamber.
  Interventions: Device: Paul glaucoma drainage device (GDD)
- GDD-tube in posterior chamber (Experimental): The Paul glaucoma drainage device consists of a plate and a tube. During surgery the plate is positioned underneath the conjunctiva and two extraocular muscles in the upper temporal or nasal quadrant of the eye. The tube is positioned in the posterior chamber.
  Interventions: Device: Paul glaucoma drainage device (GDD)

INTERVENTIONS:
Device: Paul glaucoma drainage device (GDD) — Implantation of the GDD

SUMMARY:
Rationale: Glaucoma is a group of diseases characterized by progressive neuropathy of the optic nerve associated with visual field loss. Current glaucoma management aims to preserve visual function throughout life by reducing the intraocular pressure. This can be achieved by medical therapy or by surgical procedures such as implantation of a glaucoma drainage device (GDD). Conventionally, the tube of such a device is positioned in the anterior chamber (AC). Unfortunately, the presence of the tube in the AC may have a significant negative impact on the number of endothelial cells of the cornea and may even lead to corneal decompensation. Alternatively, the tube can be positioned in the posterior chamber (i.e. behind the iris). In this study, both procedures will be compared.

Objective: Primary: to determine the loss of corneal endothelial cells after implantation of a Paul GDD with its tube either anterior or posterior of the iris. Secondary: to compare efficacy and safety of both procedures.

Study design: Prospective, randomised, treatment controlled clinical trial. Study population: Pseudophakic patients with glaucoma who need a GDD. Intervention: Implantation of a Paul GDD with its tube anterior/posterior of the iris. Main study parameters/endpoints: Endothelial cell loss of the cornea.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: At present potential benefits and drawbacks of positioning the Paul tube behind the iris are insufficiently known, successful positioning of the tube may require slightly more surgery time and the risk of hyphaema may be higher. It is expected, that in the long run damage to the corneal endothelium is less. Risks of study-related assessments are negligible, burden is low, extra time is about 35+15+35+35 minutes (total 2h).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent
* Pseudophakic
* Open angle glaucoma, pseudoexfoliation glaucoma, pigment dispersion glaucoma or angle closure glaucoma with sufficiently deep anterior chamber
* Endothelial image at baseline of fair or good quality

Exclusion Criteria:

* Iridocorneal endothelial syndrome or posterior polymorphous dystrophy
* Eyes with a history of penetrating trauma
* Eyes with a history of (intra)ocular surgery other than uncomplicated cataract surgery
* Eyes with corneal disease
* Synechiae posterior
* Pregnant and lactating women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change of endothelial cell density (ECD) | Baseline and 2 years
  ECD will be assessed at the center of the cornea and close to the tube

SECONDARY OUTCOMES:
ECD | Baseline, 6, 12 and 24 months
  ECD will be assessed at the center of the cornea and close to the tube
Intraocular pressure | Baseline, 1, 3, 6, 12 and 24 months
  Intraocular pressure
Position of the tube | Baseline, 6, 12 and 24 months
  Position of the tube on anterior segment OCT
Adverse events | Time of surgery, 1, 3, 6, 12, 24 months
  Complications at the time of surgery, postoperative adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Oogziekenhuis Rotterdam, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No